CLINICAL TRIAL: NCT01293110
Title: Database of Patients With Lower Urinary Tract Dysfunction Treated at the University of Zürich
Brief Title: Lower Urinary Tract Dysfunction Database
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Thomas Kessler, executive physician, Balgrist University Hospital
Other Study IDs: KEK-2010-0207/0/PB_2016-0189
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2024-11

CONDITIONS: Neurogenic Bladder; Diseases of the Lower Urinary Tract: General Conditions
Keywords: urodynamics; neurogenic lower urinary tract dysfunction; neurological disease/injury
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Nervous System Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with neurological disease/injury often suffer from lower urinary tract symptoms, which frequently have a negative impact on the patients' health related quality of life. The prevalence of lower urinary tract dysfunction is high and the treatment is a challenge because available treatments may fail. In this study data of patients with lower urinary tract dysfunction treated at the University of Zürich, are prospectively and systematically collected in a database.

DETAILED DESCRIPTION:
Lower urinary tract dysfunction is characterized by detrusor overactivity, detrusor sphincter dyssynergia, voiding dysfunction, stress incontinence, or a combination of these and frequently has a negative impact on the patients' health related quality of life. In addition, the treatment of lower urinary tract dysfunction is a challenge because conventional therapies may fail. Adequate treatment and long-term follow-up of lower urinary tract dysfunction is important to achieve/maintain continence and preserve renal function. Thus, we aim to prospectively collect clinical, video-urodynamic and radiological data of patients with neurogenic lower urinary tract dysfunction treated at the University of Zürich in a database.

ELIGIBILITY:
Inclusion Criteria:

* patient of Balgrist University Hospital
* patient of University Hospital Zürich
* urodynamic examination
* written informed consent

Exclusion Criteria:

* no written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ages Eligibility: minimum 18 years Genders Eligibility: female and male
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2010-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Survival of the patients | first visit to death

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Kessler, Principal Investigator — Universitätsklinik Balgrist
Locations (1):
- Spinal Cord Injury Center & Research, University of Zürich, Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walter M, Knupfer SC, Cragg JJ, Leitner L, Schneider MP, Mehnert U, Krassioukov AV, Schubert M, Curt A, Kessler TM. Prediction of autonomic dysreflexia during urodynamics: a prospective cohort study. BMC Med. 2018 Apr 13;16(1):53. doi: 10.1186/s12916-018-1040-8. PMID 29650001
- [Derived] Leitner L, Guggenbuhl-Roy S, Knupfer SC, Walter M, Schneider MP, Tornic J, Sammer U, Mehnert U, Kessler TM. More Than 15 Years of Experience with Intradetrusor OnabotulinumtoxinA Injections for Treating Refractory Neurogenic Detrusor Overactivity: Lessons to Be Learned. Eur Urol. 2016 Sep;70(3):522-8. doi: 10.1016/j.eururo.2016.03.052. Epub 2016 Apr 19. PMID 27106070